CLINICAL TRIAL: NCT02959268
Title: Pivotal Study of the Rx Al-Sense Liner for Amniotic Fluid Leakage Screening in the Second and Third Trimesters of Pregnancy
Brief Title: Pivotal Study of the Rx Al-Sense Liner for Amniotic Fluid Leakage Screening
Acronym: PRALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Common Sense (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: F-7-32.4-4
Record Dates: First submitted 2016-11-04; First posted 2016-11-09 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2017-11

CONDITIONS: Amniotic Problems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm Al-Sense diagnostic (Other): Investigator blinded to subject assessments
  Interventions: Device: Al-Sense

INTERVENTIONS:
Device: Al-Sense — Liner for diagnosis of amniotic fluid leakage verified by standard clinical diagnostic tests

SUMMARY:
This is a Prospective open-label, comparative pivotal study with comparison of self-assessments with blinded investigator assessments. Pregnant women attending the labor and delivery unit of the hospital or emergency clinic and reporting unidentified wetness (undetermined whether this is amniotic fluid leakage or urinary incontinence) will be enrolled in this study. After informed consent is obtained, each subject will be given a single AL-SENSE to use up to 12 hours or until the perception of wetness.

Product Usage

After usage, the subject will read and record any occurrence of color change of the AL-SENSE 10 minutes after the liner removal and to mark if it changes color to blue or to green or not on the designated form. The subjects will fill out the questionnaire regarding the product usage experience and the liner color reading with no help from the investigator, to validate IFU reading comprehension. A blinded clinician will perform a "standard clinical diagnosis" (clinical assessment). The standard clinical diagnostic methods will include the following tests: (1) Pooling test, (2) Ferning test, (3) pH test by pH paper. A positive Pooling test and/or positive results in both the pH test and the Ferning test will be defined as a positive clinical test result.

DETAILED DESCRIPTION:
This study is designed to demonstrate that the performance of the AL-SENSE developed by Common Sense Ltd. is safe and effective and can be used to indicate if the patient may be experiencing an amniotic fluid leakage .

The AL-SENSE is an extended shelf-life product that is technically simple, fast to react, visually readable, and therefore enables women to test the cause of any unidentified wetness, before confirmation by a physician.

Principles of operation:

Vaginal fluids are discharged over time and collected on the non-intrusive panty liner. If the user observes a blue or green stain, the result of the test is positive. The AL-SENSE polymer matrix is stained by blue or green color on a pale yellow background when the pH level of the fluid in contact with it is greater than the cutoff value.

The AL-SENSE will indicate that the pH level is elevated when the level is equal or greater than 6.5. This choice of 6.5 units as the cutoff level will limit the cases of false positive and will reduce unnecessary alarm.

Summary of Study Design

Design: Prospective open-label, comparative pivotal study with comparison of self-assessments with blinded investigator assessments.

Patient Population: Pregnant women, ages 18 and above.

Baseline/ Screening

Subjects attending the labor and delivery unit of the hospital or emergency clinic and reporting unidentified wetness (undetermined whether this is amniotic fluid leakage or urinary incontinence) will be enrolled in this study. After informed consent is obtained, each subject will be given a single AL-SENSE to use up to 12 hours or until the perception of wetness. The clinician will explain the proper use and handling of the AL-SENSE and how to read the result. The participants will be provided with instructions for use and also directed to read the Instructions For Use (IFU) prior to applying the AL-SENSE pad.

Product Usage

After usage, the subject will read and record any occurrence of color change of the AL-SENSE 10 minutes after the liner removal . The subjects will fill out the questionnaire regarding the product usage experience and the liner color reading with no help from the investigator, to validate IFU reading comprehension.

Clinical Diagnosis

A blinded clinician will perform a "standard clinical diagnosis" (clinical assessment), and record the results on a worksheet to be included in the case report form. The standard clinical diagnostic methods will include the following tests: (1) Pooling test, (2) Ferning test, (3) pH test by pH paper.

ELIGIBILITY:
Inclusion Criteria:

Screening/ Baseline inclusion criteria for subject participation in the study at baseline assessment are pregnant women age 18 and above who have completed minimum 16 weeks of pregnancy are eligible for the study. Subject attending the labor and delivery unit of the hospital or emergency clinic or outpatient clinic and reporting a feeling of vaginal wetness feeling (undetermined whether this is amniotic fluid leakage or urinary incontinence)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Color change of pantyliner surface compared to standard clinical diagnosis | 10 minutes
  Color change

SECONDARY OUTCOMES:
Questionnaire to assess subject comprehension of usage criteria and subjective experience | 15 minutes
  Self-report of product usage experience and correct usage according to instructions for use
Subject vs. Clinician reading of liner color change | up to 48 hours
  compare subject and clinician readings

CONTACTS AND LOCATIONS:
Overall Officials: Shantala Ramachandra, MD, Study Director — Consultant Medical Monitor
Locations (4):
- United States (4):
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Womens Health Institute, New Brunswick, New Jersey
  - University Hospital Rutgers Newark, Newark, New Jersey
  - Drexel University Medical School, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No